CLINICAL TRIAL: NCT03537703
Title: Transcranial Direct Current Stimulation and Effects on Early Auditory
Brief Title: Transcranial Direct Current Stimulation and Effects on Early Auditory Processing in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Walter Dunn, Staff Psychiatrist, VA Greater Los Angeles Healthcare System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: PCC 2017-080780
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Schizophrenia
Keywords: Transcranial Direct Current Stimulation; tDCS; Auditory Processing; tone matching
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Masking Description: Sham tDCS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Active tDCS + Auditory Training (Experimental): Cathodal tDCS plus concurrent active auditory training exercise
  Interventions: Combination Product: Active tDCS + Auditory Training
- Active tDCS + Control Condition (Active Comparator): Cathodal tDCS plus concurrent control condition
  Interventions: Combination Product: Active tDCS + Control Condition
- Sham tDCS + Auditory Training (Active Comparator): Sham tDCS plus concurrent active auditory training exercise
  Interventions: Combination Product: Sham tDCS + Auditory Training

INTERVENTIONS:
Combination Product: Active tDCS + Auditory Training — Active tDCS will be cathodal tDCS applied bilaterally over the auditory cortex for 20 min. The auditory training exercise will 20 min of computerized auditory training using the Sound Sweeps module of the Posit Science Brain HQ
  Arms: Active tDCS + Auditory Training
Combination Product: Active tDCS + Control Condition — Active tDCS will be cathodal tDCS applied bilaterally over the auditory cortex for 20 min. The control condition will be subjects watching a silent movie for 20 min during active tDCS stimulation.
  Arms: Active tDCS + Control Condition
Combination Product: Sham tDCS + Auditory Training — Sham tDCS will be cathodal tDCS applied bilaterally over the auditory cortex for 1 min with the current then slowly ramped down to 0 amps over the course of another minute. The auditory training exercise will 20 min of computerized auditory training using the Sound Sweeps module of the Posit Science Brain HQ
  Arms: Sham tDCS + Auditory Training

SUMMARY:
Individuals with schizophrenia have difficulties in functioning in the community. No one really knows what factors determine how well patients manage in the real world. The purpose of this pilot study is to try a new approach to improving a potential determinant of good community functioning, namely how we process sounds. Specifically, the investigators propose to examine the benefit of combining auditory training exercises with transcranial direct current stimulation (tDCS). tDCS is a new tool that is being developed as a safe and noninvasive neurostimulation method, for improving processing of sounds. Transcranial direct current stimulation involves placing a wet sponge electrode on the head and one on the arm. Electrical current from a device powered by a 9-volt battery will flow from one electrode to the other. A small portion of the current will pass through the skull and stimulate the brain. This procedure is non-invasive and painless and it results in increase or decrease of spontaneous neuronal firing in the brain. Neurons are brain cells that send electrochemical messages to each other. Its safety and beneficial effect on mental functions has been demonstrated in healthy individuals and several clinical populations. The purpose of this study is to determine if transcranial direct current stimulation added to auditory training exercises can improve how schizophrenia patients process sound.

DETAILED DESCRIPTION:
Neuroplasticity is the capacity of the brain to adapt and change in response to stimuli. In schizophrenia, structural and synaptic neuroplastic impairments potentially contribute to early perceptual processing deficits that in turn contribute to downstream higher cognitive dysfunction. The N-methyl-D-aspartate receptor (NMDA-R) hypofunction hypothesis of schizophrenia potentially explains the synaptic neuroplastic impairments as the NMDA receptor is a key component of synaptic plasticity. A rational treatment strategy involves targeting the underlying synaptic neuroplastic and perceptual processing deficits. That is, modulating the capacity for synaptic plasticity and remediating the processing deficits could then cascade into improved perceptual processing and eventually lead to better cognitive functioning.

Transcranial direct current stimulation (tDCS) is a non-invasive neurostimulation technique that has been shown to modulate synaptic plasticity. tDCS is promising because the technology is low cost and the treatment is well-tolerated and has a good safety profile. Both human and animal studies have implicated an essential role of the NMDA receptor in tDCS induced neuroplastic changes. Recent animal studies demonstrated that tDCS increased levels of an NMDA-R agonist and induced neuroplastic changes.

Cognitive training has been shown to induce both synaptic and structural neuroplastic changes in control and psychiatric patient populations. This approach targets specific neural systems with directed exercises that employ a combination of repetition, reward, and motivation to induce adaptive neuroplastic changes.

While both tDCS and cognitive training can induce synaptic plasticity changes, each approach has specific strengths that could converge in a cooperative manner. tDCS modulates NMDA-R activity and creates an environment that enhances the likelihood of synaptic changes to occur. However, tDCS alone has no inherent mechanism that drives change with specificity or directionality. Cognitive training employs targeted and repeated exercises, which confers specificity and directionality to synaptic changes. However, the extent of change that occurs is limited by the impaired state of neuroplasticity in schizophrenia. Conceivably, employing cognitive training in an environment enriched for plasticity could lead to enhanced and adaptive synaptic neuroplastic change.

Subjects who have a psychiatric illness and may be cognitively impaired will be included in the study. Persons with schizophrenia commonly have cognitive impairments that affect attention, memory, and executive functioning. There is considerable evidence that these deficits are linked to impairments in social and occupational functioning that are characteristic of the disorder.

The cognitive deficits and functional impairments of the illness are the target of interest in the study and therefore this patient population will be the specific targets for subject recruitment.

Objectives and Aims

The purpose of this proposal is to determine the effect of adding adjunctive cognitive training to tDCS in improving early auditory processing in schizophrenia patients.

Specific Aims

1. Determine if adding a cognitive auditory training exercise concurrently to cathodal tDCS offers an advantage to improving early auditory processing over tDCS alone in schizophrenia patients.
2. Determine if adding cathodal tDCS to a cognitive auditory training exercise offers an advantage to improving early auditory processing over auditory training alone in schizophrenia patients.

Study Protocol

30 individuals with schizophrenia will be randomly divided into 3 groups.

Group 1- Cathodal tDCS + auditory training exercise

Group 2- Cathodal tDCS + control condition

Group 3- Sham tDCS + auditory training exercise

Subjects in Group 1 and 2 will receive cathodal stimulation while Group 3 will receive Sham stimulation. The training component for Groups 1 and 3 will be an active auditory training program while Group 2 will engage in a control condition. On day 1, subjects will receive a baseline Tone Matching Task (TMT) and Mismatch Negativity (MMN) assessment followed by 2 sessions of tDCS. Subjects will received tDCS + training for 20 min followed by a 20 min rest period, and then a second 20 min tDCS + training session. Subjects will return the following day (approximately 21 hrs later) where they will undergo tDCS + training, a 20 min rest, and a final tDCS + training session. The post-stimulation TMT and MMN assessment will be conducted immediately following the final tDCS + training session. Each of these sessions will take approximately 3 hrs hours to complete.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-65 yrs
2. At least 3 months since any hospitalization or substantial increase in level of care for an acute exacerbation of psychotic symptoms
3. At least 6 months since any behaviors suggesting any potential danger to self or others; adherence to the regular administration of an antipsychotic medication if prescribed; dose of antipsychotic medication not varying by more than 25% over the 3 months prior to study participation;
4. Chronic medical conditions (e.g., hypertension, diabetes, dyslipidemia) consistently treated and stable for at least 3 months prior to study participation;
5. Ability to provide signed informed consent and to cooperate with study procedures.
6. Able to understand spoken English sufficiently to comprehend testing procedures

Exclusion Criteria:

1. History of treatment with electroconvulsive therapy within 6 months prior to study participation;
2. Documented history of persistent substance use disorder within 6 months prior to study participation
3. Acute medical problems
4. Metallic hardware on the scalp
5. Prior diagnosis of seizure or epilepsy
6. Subjects requiring proxy consent or consent from a legally authorized representative (LAR)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
tone matching | 40 min after last stimulation/training condition
  Performance based measure of tone discrimination

CONTACTS AND LOCATIONS:
Overall Officials: Walter Dunn, Principal Investigator — VA Medical Center-West Los Angeles
Locations (1):
- West Los Angeles VA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No